CLINICAL TRIAL: NCT00808886
Title: Comparison Between Pentacam Scheimpflug System and locs3 in Grading of Cataract
Brief Title: Study of Comparison Between Pentacam and locs3
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Soroka Medical center, Nadav Belfair, MD . Soroka Medical center
Other Study IDs: sor478308ctil
Record Dates: First submitted 2008-12-15; First posted 2008-12-16 (Estimated); Last update posted 2008-12-16 (Estimated); Status verified 2008-11

CONDITIONS: Cataract
Keywords: cataract; locs3; pentacam
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Hypothesis: There is no difference between pentacam scheimpflug system and locs3 in grading of cataract.

Major aims:

1. research the efficiency of pentacam scheimpflug system in lens density measurment.
2. To compare the pentacam with the locs3 in grading of cataract.

ELIGIBILITY:
Inclusion Criteria:

* cataract patient
* age>18

Exclusion Criteria:

* pregnant women
* any disease of the eye except for cataract
* patients who are ineligible by law to take decisions by themselves.patients who have a custodian.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: catract patients who are coming for pre- surgical evaluation.
Sampling Method: Probability Sample
Dates: Start 2008-12; Primary Completion 2009-04 (Estimated); Study Completion 2009-05 (Estimated)